CLINICAL TRIAL: NCT04235218
Title: Brief-Illness Perception Questionnaire (Brief-IPQ) Used as Prediction of Outcome in Patients With Chronic Non-malignant Pain After Six Months of Treatment in a Multidicsiplinary Pain Clinic.
Brief Title: Brief-Illness Perception Questionnaire (Brief-IPQ) Used in Patients With Chronic Non-malignant Pain.
Status: Withdrawn | Type: Observational
Why Stopped: Corona pandemic
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-081-2019
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-06

CONDITIONS: Chronic Pain Syndrome
Keywords: non-malignant pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We wish to clarify whether we can demonstrate a correlation between scores in Brief-IPQ and the effect of treatment in patients referred to our department, Interdisciplinary Pain Center Zealand University Hospital Koege, Denmark. The purpose is to outline whether we can use Brief-IPQ with Chronic Pain disorders and thereby detect those of our referred patients who are at risk for poor treatment response in an early state. In these cases, we can offer psychological intervention at the beginning of the course of treatment, in order to optimize the conditions for patients and achieve an optimal treatment effect.

DETAILED DESCRIPTION:
Chronic pain conditions are frequent in the danish population. More than 1.2 million Danes over the age of 16 are living with chronic pain. Chronic pain affects the health-related quality of life and functioning and is associated with reduced work ability, lost earnings and disability. At the Interdisciplinary Pain Center Zealand University Hospital Koege, Denmark, patients with chronic pain are received and treated based on the Bio-Psycho-Social Pain Model. The treatment of patients with complex chronic non-malignant pain can be complicated by psychological and / or social factors. The need for a screening of psychological factors in connection with the examination and planning of the pain management in the Interdisciplinary Pain Center is obvious as the patient's perception of illness and expectation of treatment have been shown to play a role in the treatment response. The Brief Illness Perception Questionnaire (Brief-IPQ) provides a quick assessment of the patient's disease perception and expectation of treatment and has proved useful in clinical practice. In this study, a Danish version of Brief-IPQ is used, which initially was taken from https://www.uib.no. Items as stated in research by L. van Oort et al (2011) have been adapted to the Danish version. A copy of the latest version can be obtained from Interdisciplinary Pain Center Zealand University Hospital Koege, Denmark.

The Study:

The study is designed as a prospective observational study of the correlation between Brief-IPQ and pain-related and demographic data in patients referred to Interdisciplinary Pain Center Zealand University Hospital Køge, Denmark. Brief IPQ and PainData (which is a database which records the well-being of Danish pain patients and operated by "Danske Regioner" and Odense University Hospital) is measured at the start of treatment and after 6 months. They will consists of items such as; Married or cohabitant, Vocational training, Educational length, Occupational status. There will furthermore be an assessment of pain type such as; nociceptive / neurogenic / generalized / visceral / other as well as the duration of symptoms and treatment with opioids: +/-, equipotent daily doses. Additionally we focus on Pain intensity (NRS) from Paindata, Psychological profile (from Paindata): anxiety, depression, stress, fear-avoidance, self-efficacy and the following changes before and after six months of treatment:

Inclusion:

All patients referred to Interdisciplinary Pain Center Zealand University Hospital Koege, Denmark and start the treatment from the start date of the study can be included in the study provided:

* Age over 18 years
* Understands and speaks Danish

Exclusion:

Patients who meet one of the following criteria are not eligible for inclusion in this study:

* Patients who do not have sufficient cognitive skills to complete the form (Brief-IPQ)
* Patients who cannot cooperate to complete the form (Brief-IPQ)
* Patients who submit invalid or illegible answers (Brief-IPQ)

Number of patients needed:

60 patients with complete data or number included as of May 1, 2020. Time schedule: Collection of data: start February 1.2020 End: when complete data has been obtained from 60 patients, or no later than 1.12.2020

Ethical aspects:

All information will be treated confidentially and all data will be anonymized by a secretary. The Investigator will keep an identification list of all patients who have been included. This list will include the patient's full name and CPR number. Collected data will be recorded in a Case Report Form. The results will be stored and analyzed using a computer and the anonymity of the patients will be preserved and local data law will be observed. Data will be stored in accordance with existing regulations. Data is stored in anonymized form and correlation and regression analysis will be performed after 6 months. The study is conducted in accordance with applicable clinical trial rules. Investigators are responsible for the handling and archiving of data in accordance with applicable rules in addition to the Act on the Processing of Personal Data and the Health Act. Data belong to the investigators. The project has been reported to the local ethic committee.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years old or older
* speak and understand written danish sufficiently to participate in the study.

Exclusion Criteria:

Patients who have insufficient cognitive abilities to answer the questions in Brief-IPQ and PainDATA. Patients who dont want to participate in the study. Patients who answer the questions in Brief-IPQ and PainDATA incompletly.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic non-malignant pain conditions reffered to the multidisciplinary pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Brief-IPQ before and after six months of treatment in a multidisciplinary pain clinic | six months
  The changes will be correlated to the following variables: pain intensity, use of opioids and self reported symptoms related to anxiety, depression, stress, fear-avoidence and self-efficacy.

SECONDARY OUTCOMES:
Influence of demographic factors on Brief-IPQ score | During the enrollment. Will be blinded to the investigators untill after the collection of data
  gener, age, education, duration of pain